CLINICAL TRIAL: NCT06680960
Title: Investigation of the Effects of Different Exercise Approaches on Exercise Capacity, Muscle Parameters and Quality of Life in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Investigation of the Effects of Different Exercise Approaches on Clinical Parameters in Chronic Obstructive Pulmonary Disease Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Cansu Özkılıçaslan, Physiotherapist, M.Sc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEŞH-BADEK-2024-553-
Record Dates: First submitted 2024-11-03; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: copd; exercise training; trunk stabilisation; muscle parameters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trunk Stabilisation Exercise Group (Active Comparator)
  Interventions: Other: Trunk stabilisation exercises
- Respiratory Exercise Group (Active Comparator)
  Interventions: Other: Respiratory exercises

INTERVENTIONS:
Other: Trunk stabilisation exercises — This exercise program includes aerobic exercise, resistance exercise and trunk stabilisation training for eight weeks.
  Arms: Trunk Stabilisation Exercise Group
Other: Respiratory exercises — This exercise program includes aerobic exercise, resistance exercise and respiratory exercise training for eight weeks.
  Arms: Respiratory Exercise Group

SUMMARY:
The beneficial effects of exercise training in individuals with chronic obstructive pulmonary disease (COPD) are well known. Standard exercise training includes structured aerobic exercise training and resistance exercise training programs applied to upper and lower extremity muscle groups. No study has been found in the literature that includes a trunk stabilization training program that includes muscles that provide whole body stabilization in COPD patients.

DETAILED DESCRIPTION:
The investigators aimed to determine the effects of an aerobic exercise training program, resistance exercise training, and an additional trunk stabilization training program in individuals with COPD.

Individuals diagnosed with COPD between the ages of 40-80 who applied to Ankara Etlik City Hospital Chest Diseases Polyclinic will be included in the study. Data collection tools and exercise training programs will be made by the same researchers. A total of 44 COPD patients, 22 in each group, will be included in the study.

COPD individuals who agree to participate in the study will be randomised electronically using a randomisation program and participants will be divided into two groups.

Group 1: Aerobic exercise training and resistance exercise training and trunk stabilisation strength training Group 2: Aerobic exercise training, resistance exercise training and respiratory exercise training

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of COPD
* Being between the ages of 40-80
* Being clinically stable (not having had an exacerbation in the last month)
* Being able to cooperate with the tests
* Not participating in any exercise training studies
* Being willing to participate in the study

Exclusion Criteria:

* Having other lung or lung involvement diseases other than COPD
* Having uncontrolled hypertension, arrhythmia and a history of myocardial infarction in the last month, unstable angina, advanced heart failure and other cardiac instability conditions
* Being hemodynamically unstable
* Being on noninvasive mechanical ventilation (NIMV) and long-term oxygen therapy (LTOT)
* Having a history of neuromuscular disease, scoliosis, chest wall surgery
* Being pregnant and having a malignancy
* Having an orthopedic or surgical problem that would prevent participation in tests and exercise training
* Not being willing to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | 8 weeks
  Maximal exercise capacity will be assessed by cardiopulmonary exercise testing (CPET) using a workload protocol of increasing intensity. Monitoring will be provided with 12-lead electrocardiography at rest, during testing and recovery. During CPET, data will be recorded with the "breathe-by-breathe" method through a face mask and a gas analyzer.

SECONDARY OUTCOMES:
Forced expiratory volume (FEV1) | 8 weeks
  It is the volume of air exhaled in the first second from the beginning of the forced vital capacity maneuver. This parameter will be assessed using spirometry (Cosmed Microquark-PC Based Spirometer, Rome, Italy) according to the criteria of the European Respiratory Society (ERS) and the American Thoracic Society (ATS). If this value is below eighty percent, it indicates the presence of airway obstruction.
Forced Vital Capacity (FVC) | 8 weeks
  It is the volume of air exhaled rapidly and forcefully following deep inspiration. Healthy people can normally exhale 80% of their lung volume in 6 seconds or less. In people with severe obstruction, this period may take up to 20 seconds. This parameter will be assessed using spirometry (Cosmed Microquark-PC Based Spirometer, Rome, Italy) according to the criteria of the European Respiratory Society (ERS) and the American Thoracic Society (ATS).
Respiratory muscle strength | 8 weeks
  Respiratory muscle strength will be assessed with a portable, electronic oral pressure measuring device (Cosmed Pony Fx, Milan, Italy). Respiratory muscle strength will be determined by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). Percentage of expected reference values according to gender and age will be used for the MIP value. The clinical significance for this patient group is 17.2 cmH2O for the measured MIP value.
COPD Assessment Questionnaire | 8 weeks
  The COPD Assessment Test (CAT) will be used to assess health status impairment in individuals with COPD. The CAT is an eight-item test consisting of questions that evaluate the severity of symptoms such as dyspnea, cough, and sputum production and the impact of the disease on daily life. It is recommended that the minimal clinical significance is a change of 2 points.
Muscle activity | 8 weeks
  Muscle activity of transversus abdominis (TrA), rectus abdominis (RA), lumbar multifidus (LM) and quadriceps muscles will be evaluated. Muscle activity will be evaluated using surface electromyography (EMG) (Neuro-MEP, Ivanovo, Russia). There is no cut-off value for these parameters in this patient group. The changes will be stated numerically and as a percentage as a result of the evaluations of the patients before and after the exercise training.
Muscle Thickness | 8 weeks
  Muscle thickness of transversus abdominis (TrA), rectus abdominis (RA), lumbar multifidus (LM) and quadriceps muscles will be evaluated. Muscle thickness will be evaluated using ultrasound (LOGIQ P9, GE Healthcare, USA). There is no cut-off value for these parameters in this patient group. The changes will be stated numerically and as a percentage as a result of the evaluations of the patients before and after the exercise training.
Timed up and go test | 8 weeks
  The Timed Up and Go Test (TUG) will be used for the balance assessment of individuals participating in the study. TUG is a frequently used, easily applicable, valid and reliable, performance-based functional mobility and balance test that evaluates dynamic balance in the clinic. It has been shown that dynamic balance impairment in COPD is associated with inadequate oxygenation and peripheral muscle weakness. Individuals who complete the test in 12 seconds or more have a risk of falling. This test, which has different cut-off values according to some disease groups, has a value of 13.5 seconds for general adults.
Functional reach test | 8 weeks
  Functional reach test will be used for the balance assessment of individuals participating in the study. Individuals who can reach 25 cm and more have a low risk of falling. Individuals who can reach between 15-25 cm have a 2 times higher risk of falling than normal. Individuals who can reach 15 cm and below have a 4 times higher risk of falling than normal. Individuals who cannot reach at all have an 8 times higher risk of falling than normal.
St George Health Questionnaire | 8 weeks
  St. George's Respiratory Questionnaire (SGRQ), a seventy-six-item health-related quality of life assessment questionnaire, will be used to assess the quality of life of the subjects.The result values are between 0 and 100 and the higher the value, the greater the degree to which the patient's quality of life is affected by the disease. Minimal significant variability in the treatment response follow-up was stated as a 4 point change.
Hospital Anxiety and Depression Scale | 8 weeks
  The Hospital Anxiety and Depression (HAD) scale will be used to determine the anxiety and depression levels of individuals participating in the study. This scale is a self-report scale that includes anxiety and depression subscales and consists of 14 items, seven of which investigate depression and seven of which investigate anxiety levels.The cut-off point for the anxiety subscale of the HAD Turkish form was found to be 10 and the cut-off point for the depression subscale was found to be 7. Patients who score above these points can be considered as a risk group. Anxiety and depression score 07: normal, 8-11: borderline, >11: anxiety and depression
Six Minute Walk Test (6MWT) | 8 weeks
  6MWT will be used to evaluate the exercise capacities of individuals who will participate in the study. The individuals' walking distance and cardiac parameters during the test will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)